CLINICAL TRIAL: NCT03142178
Title: A Double-Blind, Placebo-Controlled, Randomized Study to Evaluate the Safety and Efficacy of 3VM1001 Cream for the Treatment of Chronic Pain Caused by Osteoarthritis of the Knee: A Dose Ranging Study
Brief Title: 3VM for Treatment of Chronic Osteoarthritis Knee Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CDA Research Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3VM1216
Record Dates: First submitted 2017-04-27; First posted 2017-05-05 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2017-04

CONDITIONS: Arthritis, Degenerative
Keywords: osteoarthritis; pain; knee
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo controlled, randomized
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Experimental 3VM1001 2g X 3 daily (Experimental): 3VM1001 active cream administered 2g cream three times daily for seven days
  Interventions: Drug: Experimental: 3VM1001 active 2g Cream 3 times daily
- Placebo; 3VM1001 vehicle 2g X 3 daily (Placebo Comparator): 3VM1001 placebo vehicle administered 2g cream three times daily for seven days
  Interventions: Drug: Placebo: 3VM1001 vehicle 2g Cream 3 times daily
- Experimental 3VM1001 3g X 3 daily (Experimental): 3VM1001 active cream administered 3g cream three times daily for seven days
  Interventions: Drug: Experimental: 3VM1001 active 3g Cream 3 times daily
- Placebo; 3VM1001 vehicle 3g X3 daily (Placebo Comparator): 3VM1001 placebo vehicle administered 3g cream three times daily for seven day
  Interventions: Drug: Placebo: 3VM1001 vehicle 3g Cream 3 times daily
- Experimental 3VM1001 3g x 4 daily (Experimental): 3VM1001 active cream administered 3g cream four times daily for seven days
  Interventions: Drug: Experimental: 3VM1001 active 3g Cream 4 times daily
- Placebo; 3VM1001 vehicle 3g X 4 daily (Placebo Comparator): 3VM1001 placebo vehicle administered 3g cream four times daily for seven days
  Interventions: Drug: Placebo: 3VM1001 vehicle 3g Cream 4 times daily

INTERVENTIONS:
Drug: Experimental: 3VM1001 active 2g Cream 3 times daily — 3VM1001 2g Cream with active ingredient administered 3 times daily
  Arms: Experimental 3VM1001 2g X 3 daily
Drug: Experimental: 3VM1001 active 3g Cream 3 times daily — 3VM1001 3g Cream with active ingredient administered 3 times daily
  Arms: Experimental 3VM1001 3g X 3 daily
Drug: Experimental: 3VM1001 active 3g Cream 4 times daily — 3VM1001 3g Cream with active ingredient administered 4 times daily
  Arms: Experimental 3VM1001 3g x 4 daily
Drug: Placebo: 3VM1001 vehicle 2g Cream 3 times daily — 3VM1001 placebo 2g vehicle Cream administered 3 times daily
  Arms: Placebo; 3VM1001 vehicle 2g X 3 daily
Drug: Placebo: 3VM1001 vehicle 3g Cream 3 times daily — 3VM1001 placebo 3g vehicle Cream administered 3 times daily
  Arms: Placebo; 3VM1001 vehicle 3g X3 daily
Drug: Placebo: 3VM1001 vehicle 3g Cream 4 times daily — 3VM1001 placebo 3g vehicle Cream administered 4 times daily
  Arms: Placebo; 3VM1001 vehicle 3g X 4 daily

SUMMARY:
A double-blind, placebo-controlled, randomized dose ranging study for the use of 3VM1001 Cream, 2g three times daily, 3g three times daily, or 3g four times daily for treatment of chronic pain associated with osteoarthritis of the knee compared to inactive placebo.

DETAILED DESCRIPTION:
The study is a double-blind, placebo-controlled, dose ranging study for the use of 3VM1001 Cream, 2g three times daily, 3g three times daily, or 3g four times daily for the treatment of chronic pain associated with osteoarthritis of the knee compared to the inactive vehicle as a placebo.

A maximum of 120 subjects will be enrolled. Subjects will self-treat for 7 (+2) days, applied in the morning and at bed time.

The active pharmaceutical ingredient is copper. The proposed doses in the study are less than 2% of the upper limit of the RDA (0.9 mg/day, upper limit 10mg/day).

Rescue medication is acetaminophen, up to ~2g daily (Up to six Tylenol Regular Strength tablets).

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee according to American College of Rheumatology clinical radiological criteria. A knee radiograph will be ordered and reviewed.
* OA of the knee >/= 6 months prior to screening. Subjects with OA of both knees will treat the worst knee.
* Age 40 years or older
* Males or females of non-childbearing potential (12 or more months of spontaneous amenorrhea, bilateral oophorectomy at least 6 months prior to randomization, hysterectomy with bilateral oophorectomy at least 6 months prior to randomization, or for females over 50 years of age, hysterectomy without bilateral oophorectomy at least 6 months prior to randomization.; female subjects of childbearing potential must agree to use contraception (abstinence, birth control pills, rings or patches, diaphragm an spermicide, intrauterine device, condom and vaginal spermicide, surgical sterilization, vasectomy, progestin implant or injection); female partners of childbearing potential of male subjects must agree to use contraception as defined above.
* Moderate to severe OA pain defined a POM score between 40 mm and 90 mm.
* Baseline WOMAC pain subscale score >/=9.
* No change in physical activity and/or therapy for the past 3 months.
* All concurrent medications taken for any reason stable for 14 days
* Ability to follow protocol with reference to cognitive and situational factors such as stable housing, ability to attend visits.
* Ability to read and write English.
* Ability to apply cream without assistance.
* Able to provide written informed consent

Exclusion criteria:

* Presence of significant medical disorder that would compromise the participant's safety to take part in the study such as cancer, immunosuppressed, or evidence of alcohol or substance abuse.
* Wilson's disease or other disorder of copper metabolism.
* BMI >40
* Known hypersensitivity or allergy to any component of the product, or to acetaminophen.
* Transcutaneous electrical nerve stimulation and use of crutches, walkers or wheel chairs should be excluded prior to and during treatment. Use of a cane is permitted.
* Active conditions over the area to be treated such a eczema or psoriasis, compromised integrity of the intact, superficial skin layer over the area to be treated.
* Pain in any joint being studied that could interfere with the subject's assessment of pain in the index joint.
* Recent (within 12 months) injury (traumatic or sports related) to either knee causing pain and interference with daily activities such as walking.
* Recent (within 12 months) surgery/procedure (including intra-articular injection) to either knee causing pain that could interfere with study assessments of pain, function, and QoL.
* Extreme pain in the target knee characterized by POM score of </= 40 mm.
* Mild pain in the target knee characterized by POM score of </= 40 mm.
* Open surgery of he target knee within the last year.
* Significant concomitant disease of the knee to be studied such as fracture or osteonecrosis.
* Arthroscopic surgery of the target knee within the last 3 months.
* Use of prohibited medications/therapies during he 7-9 day treatment period including:

  1. Devices of therapeutics for knee pain or ambulation
  2. Analgesics other than acetaminpohen
  3. Systemic or locally injected corticosteroids
  4. Other investigational drugs
  5. Chemotherapy drugs
  6. Immunotherapy
  7. Topical products applied to he target knee

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Time averaged change from baseline in a standard 100 mm Visual Analog Scale (VAS). | 7 days
  The time-averaged mean of all patient pain scores over each study period.

SECONDARY OUTCOMES:
Adverse events, Serious adverse events, and study discontinuation | 8 days
  Collection of Adverse events, Serious adverse events, and study discontinuation over each study period.
Patient global impression of change scale (PGIC) from baseline to end of study period. | 8 days
  This measure is a single-item rating by participants of their improvement with treatment on a 7-point scale that ranges from "very much improved" to "very much worse" with a mid-point of "no-change".
Change in the global rating of disease for 3VM1001 Cream and placebo from baseline to the end of study. | 8 days
  Change in the global rating of disease for 3VM1001 Cream and placebo from baseline to day 8 measured on a 5-point Likert scale, with numerical values recorded by the subjects.
Patient Global Impression of change from baseline in Osteoarthritis (OA) pain.. | From screening Day 0 to the end of study (8 days)
  Subjects will rate their overall satisfaction from baseline (Day 0) to the end of study using a 6-point categorical sale from "very much worse"(0) to "very satisfied" (6).
Change in Patient Global Assessment of Treatment Satisfaction from baseline to end of study. | 8 days
  Subjects will rate their overall satisfaction with study treatment using a 5-point categorical sccale from "dissatisfied" (0) to "very satisfied" (4)
Use of rescue medication | 8 days
  The use of rescue medication for pain

CONTACTS AND LOCATIONS:
Locations (1):
- Optimed Research, LTD, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No